CLINICAL TRIAL: NCT04365569
Title: Evaluating the Effectiveness of an Individualized Nutrition and Physical Activity Counseling Program on Body Weight, Composition, Cardiovascular Function and Quality of Life in Breast Cancer Survivors
Brief Title: Evaluating the Effectiveness of an Individualized Nutrition and Physical Activity Counseling Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE11119
Record Dates: First submitted 2020-04-23; First posted 2020-04-28 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Individualized, nutrition and physical activity intervention (Experimental): Initial in-person consult with a registered dietitian, with further in-person follow-ups and monthly telephone consults
  Interventions: Behavioral: Nutrition and physical activity counseling program

INTERVENTIONS:
Behavioral: Nutrition and physical activity counseling program — 6-month interventional, counseling program based on nutrition and physical activity consisting of:
  1. Nutritional counseling by a Registered Dietitian (RD) 2) Implementation of an adequate physical activity program

SUMMARY:
More than 65% of breast cancer survivors are overweight and less than one-third participate in recommended levels of physical exercise. Obese breast cancer survivors have been found to have greater than a two-fold increase in mortality compared to women with normal body mass index (BMI). The current standard for weight loss interventions involves in-person counseling. However, this incurs costs related to travel for counseling sessions, potentially limiting program participation, compliance and sustainability.This is a pilot study of an individualized in-person and telephone-based nutrition and exercise counseling program.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer diagnosis (stage 0-III)
* Body mass index of 25mg/k2 or greater
* Actively being followed by medical oncologist, radiation oncologist, and/or breast surgeon at Maroone Cancer Center
* Able and willing to participate in nutrition counseling at Maroone Cancer Center
* Able (cleared by participant's primary oncologist) and willing to perform cardiopulmonary exercise testing
* Participants must have the ability to understand and the willingness to sign a written informed consent document
* Performance status 0 or 1 as per ECOG scale [see Appendix IV]

Exclusion Criteria:

* Body mass index below 25kg/m2
* No prior history of breast cancer
* History of metastatic disease
* Not being followed by medical oncologist, radiation oncologist, and/or breast surgeon at Maroone Cancer Center
* Unable or unwilling to participate in nutrition counseling at Maroone Cancer Center
* Participants with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Participants actively undergoing chemotherapy, immunotherapy or radiation treatment. However, participants currently taking hormonal therapy, such as selective estrogen receptor modulators (SERMS), or aromatase inhibitors, may be included in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2024-05-16 (Actual)

PRIMARY OUTCOMES:
Percent of participants achieving 10% weight loss | At baseline
  Efficacy of intervention as assessed by percent of participants achieving 10% weight loss
Percent of participants achieving 10% weight loss | At 3 months
  Efficacy of intervention as assessed by percent of participants achieving 10% weight loss
Percent of participants achieving 10% weight loss | At 6 months
  Efficacy of intervention as assessed by percent of participants achieving 10% weight loss
Compliance to the recommended dietary pattern | At 3 months
  Assess compliance to the recommended dietary pattern, diet quality scores will be calculated by the RD after monthly telephone consults or in-person at 3 months and 6 months into the intervention. Each of the 3 elements will be scored from 0-3, resulting in a total score range from 0-9
Compliance to physical activity goal | At 6 months
  Percent of participants complying with proposed activity goal of 150 minutes of moderate intensity physical activity or 75 minutes of vigerous intensity physical activity (or a combination of both) per week over six months

SECONDARY OUTCOMES:
Body fat percentage | Baseline
  Body fat percentage measured by the registered dietitian (RD) using bioelectrical impedance analysis
Body fat percentage | 3 months
  Body fat percentage measured by the registered dietitian (RD) using bioelectrical impedance analysis
Body fat percentage | 6 months
  Body fat percentage measured by the registered dietitian (RD) using bioelectrical impedance analysis
Glycemic control as measured by HbA1c | At 3 months
  Glycemic control as measured by HbA1c
Glycemic control as measured by HbA1c | At 6 months
  Glycemic control as measured by HbA1c
Cholesterol | At 3 months
  Effect of the intervention on lipid profile as measured by high density cholesterol levels
Cholesterol | At 6 months
  Effect of the intervention on lipid profile as measured by high density cholesterol levels
Low density lipoprotein | At 3 months
  Effect of the intervention on lipid profile as measured by low density lipoprotein levels
Low density lipoprotein | At 6 months
  Effect of the intervention on lipid profile as measured by low density lipoprotein levels
high density lipoprotein | At 3 months
  Effect of the intervention on lipid profile as measured by high density lipoprotein levels
high density lipoprotein | At 6 months
  Effect of the intervention on lipid profile as measured by high density lipoprotein levels
Triglycerides | At 3 months
  Effect of the intervention on lipid profile as measured by triglyceride levels
Triglycerides | At 6 months
  Effect of the intervention on lipid profile as measured by triglyceride levels
Serum vitamin D | At 3 months
  Effect of the intervention on serum vitamin D
Serum vitamin D | At 6 months
  Effect of the intervention on serum vitamin D
Serum C-reactive protein (CRP) | At 3 months
  Effect of the intervention on CRP
Serum C-reactive protein (CRP) | At 6 months
  Effect of the intervention on CRP
Maximum oxygen uptake as measured by VO2 max | Baseline
  Maximum oxygen uptake as measured by VO2 max
Maximum oxygen uptake as measured by VO2 max | At 3 months
  Maximum oxygen uptake as measured by VO2 max
Maximum oxygen uptake as measured by VO2 max | At 6 months
  Maximum oxygen uptake as measured by VO2 max

OTHER OUTCOMES:
Quality of life as measured by Functional Assessment of Cancer Therapy - Breast Cancer (FACT-B) | Baseline, 3 months and 6 months
  Quality of life as measured by Functional Assessment of Cancer Therapy - Breast Cancer (FACT-B), a 36-item self-report questionnaire to assess the quality of life as reported by breast cancer survivors with scores ranging from 0 to 123, and lower scores indicating better health.
Quality of life as measured by Brief Pain Inventory (BPI) | Baseline, 3 months and 6 months
  Quality of life as measured by Brief Pain Inventory (BPI), a 9-item self-administered questionnaire that can evaluate the effect of an individual's pain on their daily functioning. This is a 10-point scale with 0 being the best possible score, meaning "no pain", and 10 being the worst possible score, meaning "pain as bad as you can imagine"
Quality of life as measured by Generalized Anxiety Disorder-7 (GAD-7) | Baseline, 3 months and 6 months
  Quality of life as measured by Generalized Anxiety Disorder-7 (GAD-7), a 7-item self-report questionnaire measuring anxiety which uses a four-point rating scale (ranging from 0 to 3) asking how often in the last two weeks participants have experienced symptoms pertaining to feeling anxious, worried, difficulty relaxing, and irritability. Higher scores indicate higher distress. with a possible score range of 0 to 21 with higher scores indicating worse anxiety.
Quality of life as measured by Patient Health Questionnaire-9 (PHQ-9) | Baseline, 3 months and 6 months
  Quality of life as measured by Patient Health Questionnaire-9 (PHQ-9), which objectifies degree of depression severity with a possible score range of 0 to 27 and higher scores indicating worse outcomes
Quality of life as measured by NCCN Distress Thermometer | Baseline, 3 months and 6 months
  Quality of life as measured by NCCN Distress Thermometer, which measures distress on a scale of 0 to 10, with higher scores indicating worse distress
Factors associated with adherence to the program | At 6 months
  Factors to be assessed include age, race, time since diagnosis, time since last chemotherapy, medical comorbidities and other lifestyle factors such as alcohol consumption and smoking

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Stone, MD, Principal Investigator — Cleveland Clinic, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Florida Weston, Case Comprehensive Cancer Center, Weston, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Will share IPD with other researchers within the same institution, but not outside the institution
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code